CLINICAL TRIAL: NCT02772627
Title: A Double-blind, Randomised, Placebo-controlled, Rising Multiple Dose Study to Investigate the Tolerability, Steady-state Pharmacokinetics and Erythrocyte COMT Inhibition of BIA 3-202 in Healthy Volunteers.
Brief Title: Study to Investigate the Tolerability, Steady-state Pharmacokinetics and Erythrocyte COMT Inhibition of BIA 3-202
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-3202-105
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, Nebicapone
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nebicapone 100 mg / Placebo (Experimental): Treatment consisted of nebicapone/placebo repeated administration: one dose at 4-h intervals, for 7 full days: first dose at approximately 08 h (±1 h) on Day 1 and final dose at approximately 08 h (±1 h) on Day 8. Within each group (n=8), 2 volunteers were be randomised to receive placebo and the remaining 6 volunteers to receive nebicapone.
  Interventions: Drug: Nebicapone; Drug: Placebo
- Nebicapone 200 mg / Placebo (Experimental): Treatment consisted of nebicapone/placebo repeated administration: one dose at 4-h intervals, for 7 full days: first dose at approximately 08 h (±1 h) on Day 1 and final dose at approximately 08 h (±1 h) on Day 8. Within each group (n=8), 2 volunteers were be randomised to receive placebo and the remaining 6 volunteers to receive nebicapone.
  Interventions: Drug: Nebicapone; Drug: Placebo
- Nebicapone 300 mg / Placebo (Experimental): Treatment consisted of nebicapone/placebo repeated administration: one dose at 4-h intervals, for 7 full days: first dose at approximately 08 h (±1 h) on Day 1 and final dose at approximately 08 h (±1 h) on Day 8. Within each group (n=8), 2 volunteers were be randomised to receive placebo and the remaining 6 volunteers to receive nebicapone.
  Interventions: Drug: Nebicapone; Drug: Placebo

INTERVENTIONS:
Drug: Nebicapone — Nebicapone 100 mg tablets; oral route.
  Other Names: BIA 3-202
Drug: Placebo — Placebo tablets; oral route.

SUMMARY:
The purpose of this study is to investigate the tolerability and safety of three multiple dose regimens of nebicapone (BIA 3-202 100 mg, 200 mg, and 300 mg 6 times daily) in healthy volunteers. To characterise the steady-state pharmacokinetic and erythrocyte COMT inhibition profiles of nebicapone in healthy volunteers.

DETAILED DESCRIPTION:
Study design and methodology:

This was a single centre, human pharmacology (phase I), double-blind, randomised, placebo-controlled study of three multiple rising doses in three sequential groups of healthy volunteers. Subjects were screened for eligibility within 28 days of admission.

Screening:

Screening consisted of review of medical history, physical examination, neurological examination, vital signs, 12-lead ECG, clinical laboratory safety tests (haematology, coagulation, plasma biochemistry, urinalysis, HBsAg, anti-HCV Ab, anti-HIV-1 and anti-HIV-2 Ab), drugs of abuse and alcohol screen, and written informed consent. A pregnancy test was performed in all female subjects. The investigator was informed of the screening results prior to the subject's admission.

Treatment period:

Eligible subjects were admitted to the UFH for one treatment period on the morning of the day prior to receiving the first dose of trial medication and remained in the UFH until at least 48 hours after receiving their final dose of trial medication (final dose: Day 8; leaving the UFH: Day 10). Then, they were to leave and to return on the Days 15, 22 and 29 for the 168 h, 336 h, and 504 h post final dose blood samples and clinical evaluations. Trial medication was administered at 4-h intervals (Group 1: Nebicapone 100 mg/Placebo, 6 times/day; Group 2: Nebicapone 200 mg/Placebo, 6 times/day; Group 3: Nebicapone 300 mg/Placebo, 6 times/day).

On admission (Day -1), subjects had a physical examination, medical history update, vital signs (blood pressure and heart rate), neurological examination, 12-lead ECG, clinical laboratory tests (haematology, coagulation, plasma biochemistry, urinalysis), pregnancy test, screen for drugs of abuse and alcohol, and 24-h urine collection for the assay of urinary electrolytes and creatinine.

On Day 1, Nebicapone /Placebo started being administered at 4 hourly intervals, until the final dose on Day 8.

The following assessments were performed as described: vital signs (blood pressure and heart rate) at Days 1 to 7 pre and 1 hour post 08, 12, 16, 20 and 24 h doses, and Day 8 pre-dose and 1, 24, 48, 168, 336 hours post final dose, and at Day 29; physical examination: admission, at Day 10 and Day 29; neurological examination at on admission, pre-dose and 2 hours post 08, 12, 16, 20 and 24 h doses on Day 1, 2 hours post 08h00 and 20h00 doses on Days 2 to 7, and 2 hours post 08h00 dose on Day 8; 12-lead ECG at 1 hour post 08h00 dose on Days 1, 2, 3, 5 and 8, and 48 h post final dose, and Day 29; continuous lead-II ECG monitoring at 0-6 hours post first dose on Day 1, and 0-4 hours post 08h00 dose on Day 8; blood samples (7 ml) for the assay of plasma nebicapone and its metabolites, and for the assay of the erythrocyte soluble COMT (S-COMT) activity were taken at Day 1, pre-dose, ½, 1, 1½, 2, 3, 4, 8, 12 and 16 hours post first dose (08h00), at Day 8, pre final dose (08h00), ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 168*, 336*, and 504* hours post final dose (*only for the assay of plasma nebicapone metabolites), and at Days 2, 3, 4, 5, 6, and 7, pre 08h00 and 20h00 doses; urine and blood collection for urinalysis, coagulation, haematology and plasma biochemistry at admission, and on Days 2, 10 and 29; and 24-h urine collection for the assay of urinary electrolytes and creatinine at admission, and on Days 1 and 9.

Adverse events were monitored throughout.

Follow-up:

The end-of-study assessments took place after the last blood sample (504 h) and included: medical history review, physical examination, vital signs, 12-lead ECG, clinical laboratory safety tests, adverse events; pregnancy test (if female).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive.
* Subjects who were healthy as determined by pre study medical history, physical examination, and 12- lead ECG.
* Subjects who had clinical laboratory tests acceptable to the investigator.
* Subjects who were negative for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for drugs of abuse and alcohol at screening and admission.
* Subjects who were non-smokers or who smoke less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, or
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had an acute infection such as influenza at the time of screening and/or admission.
* Subjects who had used prescription drugs within 4 weeks of first dosing.
* Subjects who had used oral contraceptives or over the counter medication excluding oral routine vitamins but including mega dose vitamin therapy within one week of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of their first admission to this study.
* Subjects who had previously received BIA 3-202.
* Subjects who had donated and/or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans and/or have medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method or she used oral contraceptives.
* Subjects who were unwilling or unable to give written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2001-09; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) - Nebicapone | Day 8
  Mean nebicapone plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)
Time of maximum observed concentration (tmax) - Nebicapone | Day 8
  Mean nebicapone plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)
Area under the plasma concentration time curve extrapolated to infinity (AUC0-∞) - Nebicapone | Day 8
  Mean nebicapone plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)
Apparent terminal elimination half-life (t1/2) - Nebicapone | Day 8
  Mean nebicapone plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)
Maximum observed plasma concentration (Cmax) - 3-O-methylnebicapone (BIA 3-270) | Day 8
  Mean 3-O-methylnebicapone (BIA 3-270) plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)
Time of maximum observed concentration (tmax) - 3-O-methylnebicapone (BIA 3-270) | Day 8
  Mean 3-O-methylnebicapone (BIA 3-270) plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)
Area under the plasma concentration time curve extrapolated to infinity (AUC0-∞) - 3-O-methylnebicapone (BIA 3-270) | Day 8
  Mean 3-O-methylnebicapone (BIA 3-270) plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)
Apparent terminal elimination half-life (t1/2) - 3-O-methylnebicapone (BIA 3-270) | Day 8
  Mean 3-O-methylnebicapone (BIA 3-270) plasma concentration-time profiles following the last dose (Day 8) of a multiple-dose oral administration of nebicapone (100 mg, 200 mg or 300 mg, at 4-h intervals)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit - BIAL - Portela & Ca, S.A., S. Mamede Do Coronado, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: No